CLINICAL TRIAL: NCT03203694
Title: Restoring Vasodilator Actions of Insulin in Patients With Type 2 Diabetes
Brief Title: Effects of Walking and Heating on Vascular Function in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jaume Padilla, Associate Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008181
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a walking, a lower body heating, or no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Walking: Intervention arm in diabetics (Experimental): The walking program will consist of 45 minutes of walking (at a moderate pace) 5 days per week for 8 weeks.
  Interventions: Behavioral: Walking: Intervention arm in diabetics
- Walking: No intervention in diabetics (Experimental): Subjects will be instructed to continue their usual lifestyle for 8 weeks.
  Interventions: Other: Walking: No intervention in diabetics
- Walking: Healthy cohort as reference controls (Other): Subjects will be studied at one time only.
  Interventions: Other: Walking: Healthy cohort as reference controls
- Lower body heating: Intervention arm in healthy subjects (Experimental): This intervention consists of 60 minutes of lower body heating (40-42 degree C).
  Interventions: Behavioral: Lower body heating: Intervention arm in healthy subjects
- Lower body heating: Intervention arm in diabetics (Experimental): This intervention consists of 60 minutes of lower body heating (40-42 degree C) 7 days per week for 7 days.
  Interventions: Behavioral: Lower body heating: Intervention arm in diabetics
- Lower body heating: Healthy cohort as reference controls (Other): Subjects will be studied at one time only.
  Interventions: Other: Lower body heating: Healthy cohort as reference controls

INTERVENTIONS:
Behavioral: Walking: Intervention arm in diabetics — The walking program will consist of 45 minutes of walking (at a moderate pace) 5 days per week for 8 weeks.
  Arms: Walking: Intervention arm in diabetics
Other: Walking: No intervention in diabetics — Subjects will be instructed to continue their usual lifestyle for 8 weeks.
  Arms: Walking: No intervention in diabetics
Other: Walking: Healthy cohort as reference controls — Subjects will be studied at one time only.
  Arms: Walking: Healthy cohort as reference controls
Behavioral: Lower body heating: Intervention arm in healthy subjects — This intervention consists of 60 minutes of lower body heating (40-42 degree C).
  Arms: Lower body heating: Intervention arm in healthy subjects
Behavioral: Lower body heating: Intervention arm in diabetics — This intervention consists of 60 minutes of lower body heating (40-42 degree C) 7 days per week for 7 days.
  Arms: Lower body heating: Intervention arm in diabetics
Other: Lower body heating: Healthy cohort as reference controls — Subjects will be studied at one time only.
  Arms: Lower body heating: Healthy cohort as reference controls

SUMMARY:
The purpose of the present study is to determine the effects of increased walking and lower body heating on leg vascular function in patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The notion that habitual aerobic exercise increases insulin-induced vasodilation is largely founded on rodent studies, hence the urgent need for human studies, especially in patients with type 2 diabetes (T2D). For example, it remains unknown if increased walking, the most common form of physical activity, enhances skeletal muscle vasodilator actions of insulin in T2D. In addition, the molecular mechanisms by which exercise improves vasoreactivity to insulin have not been examined in humans. The investigators propose that in T2D patients who are sedentary (i.e., the vast majority), increased leg blood flow with walking or local heating signifies a vital strategy to correct vascular insulin resistance. This study will establish whether increased physical activity and associated hemodynamic forces (e.g., shear stress) are a direct form of vascular medicine in humans.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes who are overweight and obese (BMI 25-50 kg/m2), 35 to 65 years of age, and sedentary (<60 minutes structured exercise/week). Healthy volunteers without type 2 diabetes: 18 to 65 years of age.

Exclusion Criteria:

1. Cardiovascular disease including myocardial infraction, heart failure, coronary artery disease, stroke;
2. renal or hepatic diseases;
3. active cancer;
4. autoimmune diseases;
5. immunosuppressant therapy;
6. excessive alcohol consumption (>14 drinks/week for men; >7 drinks/week for women);
7. current tobacco use;
8. pregnancy;
9. mobility limitations;
10. foot ulcers;
11. diabetic neuropathy
12. uncontrolled hypertension (>=180 systolic / 100 diastolic mmHg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Padilla, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Walking: Intervention Arm in Diabetics | Walking: No Intervention in Diabetics | Walking: Healthy Cohort as Reference Controls | Lower Body Heating: Intervention Arm in Healthy Subjects | Lower Body Heating: Intervention Arm in Diabetics | Lower Body Heating: Healthy Cohort as Reference Controls
Started | 13 | 13 | 15 | 18 | 20 | 20
Completed | 11 | 13 | 15 | 18 | 20 | 20
Not Completed | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking: Intervention Arm in Diabetics | Walking: No Intervention in Diabetics | Walking: Healthy Cohort as Reference Controls | Lower Body Heating: Intervention Arm in Healthy Subjects | Lower Body Heating: Intervention Arm in Diabetics | Lower Body Heating: Healthy Cohort as Reference Controls | Total
Number analyzed (Participants) | 13 | 13 | 15 | 18 | 20 | 20 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 15 | 18 | 20 | 20 | 99
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 10 | 8 | 12 | 12 | 54
  Male | 7 | 7 | 5 | 10 | 8 | 8 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4 | 0 | 4 | 12
  Not Hispanic or Latino | 12 | 13 | 12 | 14 | 20 | 16 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 5 | 0 | 7
  White | 13 | 12 | 15 | 17 | 15 | 20 | 92
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 15 | 18 | 20 | 20 | 99
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Drop out subjects are not included in the BMI calculation.
  kg/m^2
    number analyzed (Participants) | 11 | 13 | 15 | 18 | 20 | 20 | 97
    (all) | 36.9 (1.6) | 36.2 (1.7) | 23.5 (2.3) | 25.1 (4.2) | 35.9 (1.2) | 23.7 (2.2) | 29.6 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Insulin-stimulated Leg Blood Flow Calculated as Percent Change (t0, t60)
Description: Measure of blood flow in response to insulin. Blood flow is measured via Doppler ultrasound at the femoral artery. Measurements are performed at baseline (t0) and after 60 minutes of insulin stimulation (t60).
Time Frame: Percent change from baseline leg blood flow during 60 minutes of insulin stimulation.
Population: Outcomes data from participants who were assigned to an intervention arm are reported under Outcome 2 (change from baseline to post-intervention).
Measure: Mean (Standard Error); unit: percentage change
Groups:
- Experimental: Lower Body Heating: Intervention Arm in Diabetics: This intervention consists of 60 minutes of lower body heating (40-42 degree C) 7 days per week for 7 days.
Arm/Group | Walking: Intervention Arm in Diabetics | Walking: No Intervention in Diabetics | Walking: Healthy Cohort as Reference Controls | Lower Body Heating: Intervention Arm in Healthy Subjects | Experimental: Lower Body Heating: Intervention Arm in Diabetics | Lower Body Heating: Healthy Cohort as Reference Controls
Number analyzed (Participants) | 0 | 0 | 15 | 0 | 0 | 20
percentage change |  |  | 133.6 (48.7) |  |  | 8.92 (2.26)

2. Primary Outcome: Net Change in Insulin-stimulated Leg Blood Flow Calculated as Percent Change From Pre-intervention (t0,t60) to Post-intervention (t0,t60).
Description: Measure of blood flow in response to insulin. Blood flow is measured via Doppler ultrasound at the femoral artery. Measurements are performed pre-intervention and post-intervention at baseline (t0) and after 60 minutes of insulin stimulation (t60). Outcome measure indicates whether percent change in insulin-stimulated blood flow increased or decreased following intervention. Interventions that show an increase demonstrate an improvement in insulin-stimulated blood flow.
Time Frame: Change from baseline insulin-stimulated leg blood flow following 1 heating session, 7 days of heating intervention, or 8 weeks of walking intervention/no intervention.
Population: Outcomes data from participants who were not assigned a treatment arm are reported under Outcome 1 (Percent change in insulin-stimulated blood flow).
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Walking: Intervention Arm in Diabetics | Walking: No Intervention in Diabetics | Walking: Healthy Cohort as Reference Controls | Lower Body Heating: Intervention Arm in Healthy Subjects | Lower Body Heating: Intervention Arm in Diabetics | Lower Body Heating: Healthy Cohort as Reference Controls
Number analyzed (Participants) | 11 | 13 | 0 | 18 | 20 | 0
percent change | 15.9 (47.3) | -17.6 (21.4) |  | 60.2 (18.5) | 11.1 (3.5) |

ADVERSE EVENTS:
Time Frame: 8 weeks: (Walking: Intervention arm in diabetics; Walking: No intervention in diabetics) 7 days: (Lower body heating: Intervention arm in healthy subjects; Lower body heating: Intervention arm in diabetics) 1 day (1 session): (Walking: Healthy cohort as reference controls; Lower body heating: Healthy cohort as reference controls)
Arm/Group | Walking: Intervention Arm in Diabetics | Walking: No Intervention in Diabetics | Walking: Healthy Cohort as Reference Controls | Lower Body Heating: Intervention Arm in Healthy Subjects | Lower Body Heating: Intervention Arm in Diabetics | Lower Body Heating: Healthy Cohort as Reference Controls
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/15 | 0/18 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/15 | 0/18 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/13 | 0/13 | 0/15 | 1/18 | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Walking: Intervention Arm in Diabetics (N=13) | Walking: No Intervention in Diabetics (N=13) | Walking: Healthy Cohort as Reference Controls (N=15) | Lower Body Heating: Intervention Arm in Healthy Subjects (N=18) | Lower Body Heating: Intervention Arm in Diabetics (N=20) | Lower Body Heating: Healthy Cohort as Reference Controls (N=20)
Allergic response to contrast agent (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Experience of allergic skin reaction to Definity (Perflutren) contrast agent.
Vasovegal Reaction (Vascular disorders) | 0 (0) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Vaso-vegal reaction in response to IV placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03203694/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03203694/SAP_001.pdf
  • Informed Consent Form: Lower body heating (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT03203694/ICF_002.pdf
  • Informed Consent Form: Lower body heating: Healthy cohort as reference controls (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT03203694/ICF_003.pdf
  • Informed Consent Form: Walking (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT03203694/ICF_004.pdf